CLINICAL TRIAL: NCT06663085
Title: The Effect of Enteral Feeding on Splanchnic Oxygenation During Blood Transfusion in Preterm Infants
Brief Title: Using NIRS to Evaluate Splanchnic Oxygenation During Blood Transfusion in Preterm Infant
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gadjah Mada University (Other)
Responsible Party: Principal Investigator, Leksmana Hidayatullah, MD, Gadjah Mada University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: KE/FK/1583/EC/2024
Record Dates: First submitted 2024-10-24; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Splanchnic Oxygenation; NIRS; PreTerm Neonate; Enteral Feeds
Keywords: transfusion; nirs; splanchnic oxygenation; preterm neonate; enteral feeds
MeSH Terms: interventions — Enteral Nutrition

STUDY DESIGN:
Intervention Model Description: control group: not received enteral feeding during transfusion intervention group: received enteral feeding
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group not received enteral feeding (No Intervention): control group not received enteral feeding during blood transfusion
- intervention group received enteral feeding (Active Comparator): intervention group still received enteral feeding during blood transfusion
  Interventions: Dietary Supplement: Enteral feeding

INTERVENTIONS:
Dietary Supplement: Enteral feeding — intervention group received enteral feeding breastmilk during transfusion
  Other Names: breastmilk
  Arms: intervention group received enteral feeding

SUMMARY:
To evaluate the differences splanchnic oxygen saturation in preterm infants receiving red blood cell transfusion with and without enteral feeding, and their outcomes.

DETAILED DESCRIPTION:
using NIRS to evaluate splanchnic oxygenation

ELIGIBILITY:
Inclusion Criteria:

* Infant with gestational age < 37 weeks
* Planned to receive blood transfusion
* Had received minimum 25 ml/kg/day enteral feeding
* in stable condition

Exclusion Criteria:

* Infant with multiple congenital anomalies
* Infant with suspected/confirmed genetic anomalies
* Parents or family did not sign the informed consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-10-30 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
cerebral splanchnic oxygenation ratio using nirs | from enrollment to 48 hours after transfusion
  percentage of splanchnic oxygenaation divided with cerebral oxygenation

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Sardjito General Hospital, Yogyakarta, Special Region of Yogyakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No
the data will not be planned to share until publication, if any person want to see the data can contact the investigator by email